CLINICAL TRIAL: NCT06785818
Title: A Registry to Assess Long-Term Safety of Patients With B-Lymphocyte Malignancies Treated With Tisagenlecleucel in South Korea
Brief Title: Long-term Follow up Local Registry Study of Kymriah in South Korea
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019CKR02
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: B-Cell Acute Lymphoblastic Leukemia, Diffuse Large B-Cell Lymphoma, Follicular Lymphoma
Keywords: B-Lymphocyte Malignancies; B-ALL; DLBCL; FL; Tisagenlecleucel; South Korea
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — tisagenlecleucel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tisagenlecleucel: Patients who have been treated with tisagenlecleucel
  Interventions: Other: Tisagenlecleucel

INTERVENTIONS:
Other: Tisagenlecleucel — This is an observational study. There is no treatment allocation. The decision to initiate tisagenlecleucel will be based solely on clinical judgement.
  Other Names: Kymriah®

SUMMARY:
This study is multicenter, primary data collection, non-interventional registry study to assess long-term safety, secondary malignancy risk, and effectiveness of tisagenlecleucel in patients with B-cell malignancies in a routine clinical practice setting in Korea.

DETAILED DESCRIPTION:
This study will inform on long-term real-world safety and effectiveness of tisagenlecleucel. The primary objective is to evaluate the long-term safety and the risk of secondary malignancies in patients with B lymphocyte malignancies treated with tisagenlecleucel in a real-world setting. The main secondary objective is to evaluate the longterm effectiveness of tisagenlecleucel.

All participants enrolled in this study will be followed up for 15 years from the time of Kymriah® infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who receive tisagenlecleucel infusion in the commercial setting, treated under a managed access program or other pathway, e.g., when product was manufactured for the commercial setting but turned out to be out of specification (OOS).
2. Consented to data collection.

Exclusion Criteria:

1. Patients who are enrolled or will be enrolled in the Novartis long term follow-up protocol CCTL019A2205B.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with B-Lymphocyte Malignancies Treated with Tisagenlecleucel in South Korea
Sampling Method: Non-Probability Sample
Enrollment: 179 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2039-12-30 (Estimated); Study Completion 2039-12-30 (Estimated)

PRIMARY OUTCOMES:
The type and frequency of AEs, ADRs, SAEs, SADRs, UAEs, UADRs, USAEs, USADRs, AESI | Up to 15 years post-infusion
  The type and frequency of adverse event (AE)/adverse drug reaction (ADR)/ serious adverse event (SAE)/serious adverse drug reaction (SADR)/ unexpected adverse event (UAE)/unexpected adverse drug reaction (UADR)/ unexpected serious adverse event (USAE)/unexpected serious adverse drug reaction (USADR)/ adverse event of special interest (AESI)
Identify participants for chimeric antigen receptor (CAR) transgene detection and/or CAR surface expression (if applicable). | Up to 15 years post-infusion
  When applicable, identify patients for CAR transgene detection and/or CAR surface expression by quantitative polymerase chain reaction (q-PCR), in-situ hybridization, flow cytometry and/or immunohistochemistry (IHC), whichever testing is appropriate, in relevant samples (blood, bone marrow, etc.)
Identify presence of replication competent lentivirus (RCL) in blood or tissues | Up to 15 years post-infusion
  Replication competent lentiviruses (RCL) are virus particles capable of infecting cells and replicating to produce additional infectious particles.

SECONDARY OUTCOMES:
B-Cell Acute Lymphoblastic Leukemia - Overall response rate (ORR) | Up to 15 years post-infusion
  The overall response rate (ORR) is defined as the percentage of subjects with a best overall disease response of complete response (CR) or Complete remission with incomplete blood count recovery (CRi). For ALL (Acute Lymphoblastic Leukemia), complete remission is defined as: less than 5% blasts in marrow, less than 1% blasts in blood and no EM disease.
B-Cell Acute Lymphoblastic Leukemia - Duration of response (DOR) | Up to 15 years post-infusion
  Duration of Response (DoR) is defined as the time from first documented evidence of response (the first response prior to confirmation) until time of documented disease progression or death due to any cause, whichever was first.
B-Cell Acute Lymphoblastic Leukemia - Relapse-free survival (RFS) | Up to 15 years post-infusion
  RFS is defined as the time from the date of first dose of the study treatment to the date of the first documented disease recurrence or death due to any cause whichever comes first.
B-Cell Acute Lymphoblastic Leukemia - Event-free survival (EFS) | Up to 15 years post-infusion
  Event free survival is the time from the date of start of treatment to the earliest of the following:
  * Death from any cause after remission
  * Relapse
  * Treatment failure (failure to achieve remission, including death without remission)
B-Cell Acute Lymphoblastic Leukemia - Proportion of patients with minimal residual disease (MRD) negative status in bone marrow who achieve a best overall response (BOR) of CR or CRi | Up to 15 years post-infusion
  MRD is a term used to describe a very small number of cancer cells that remain in the body during or after treatment. MRD is defined as positive by immunophenotype if 1/1000 cells is positive.
Diffuse Large B-Cell Lymphoma - Overall response rate (ORR) | Up to 15 years post-infusion
  The overall response rate (ORR) is defined as the percentage of subjects with a best overall disease response of complete response (CR) or Partial response (PR)
Diffuse Large B-Cell Lymphoma - DOR | Up to 15 years post-infusion
  Duration of Response (DoR) is defined as the time from first documented evidence of response (the first response prior to confirmation) until time of documented disease progression or death due to any cause, whichever was first.
Diffuse Large B-Cell Lymphoma - RFS | Up to 15 years post-infusion
  RFS is defined as the time from the date of first dose of the study treatment to the date of the first documented disease recurrence or death due to any cause whichever comes first.
Diffuse Large B-Cell Lymphoma - Progression-free survival (PFS) | Up to 15 years post-infusion
  Progression-free survival is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause whichever comes first.
Diffuse Large B-Cell Lymphoma - Overall survival (OS) | Up to 15 years post-infusion
  Overall survival is the time from date of start of treatment to the date of death due to any reason.
Follicular Lymphoma - ORR | Up to 15 years post-infusion
  The overall response rate (ORR) is defined as the percentage of subjects with a best overall disease response of complete response (CR) or Partial response (PR)
Follicular Lymphoma -Complete response rate (CRR) | Up to 15 years post-infusion
  Complete response rate is the proportion of patients with a complete disease response, which is defined as the best disease response recorded from date of start of treatment until progressive disease or start of new anticancer therapy, whichever comes first.
Follicular Lymphoma - DOR | Up to 15 years post-infusion
  Duration of Response (DoR) is defined as the time from first documented evidence of response (the first response prior to confirmation) until time of documented disease progression or death due to any cause, whichever was first.
Follicular Lymphoma - RFS | Up to 15 years post-infusion
  RFS is defined as the time from the date of first dose of the study treatment to the date of the first documented disease recurrence or death due to any cause whichever comes first.
Follicular Lymphoma - PFS | Up to 15 years post-infusion
  Progression-free survival is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause whichever comes first.
Follicular Lymphoma - Overall survival (OS) | Up to 15 years post-infusion
  Overall survival is the time from date of start of treatment to the date of death due to any reason.
Frequency and rate of pregnancy outcomes | Up to 15 years post-infusion
  pregnancy outcomes:
  * Live birth, at term (presence or absence of congenital abnormality)
  * Live birth, premature (presence or absence of congenital abnormality)
  * Intrauterine fetal death
  * Spontaneous abortion
  * Elective abortion
  * Unknown

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- South Korea (8):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Incheon, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul

IPD SHARING:
Plan to Share IPD: No